CLINICAL TRIAL: NCT05400109
Title: A Phase 1/1b Multicenter, Open Label Study to Evaluate the Safety of UF-KURE19 Cells in Patients With B Cell Non-Hodgkin Lymphomas
Brief Title: Evaluate the Safety of UF-KURE19 Cells in Non-Hodgkin Lymphomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Wald (Other)
Responsible Party: Sponsor-Investigator, David Wald, IND Holder, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2422
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Non Hodgkin Lymphoma
Keywords: UF-KURE19; CD19 CAR-T cells; Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- UF-KURE19 CAR-T cell infusion (Experimental): The safety and manufacturing feasibility of UF-KURE19 will be determined with up to 10 patients being enrolled. Lymphodepleting therapy will begin on Days -4 to -2 with each weight category of participants receiving 30mg/m2/IV of Fludarabine and 500mg/m2/IV of Cyclophosphamide regardless of the level of UF-KURE19 CAR-T cell dosing.
  Dosing:
  Participants greater than or equal to 50 kg:
  * Level -1: 10 x 10^6 UF-KURE19 CAR-T Cell Dose (CAR positive cells)
  * Level 1 : 17.5 x 10^6 UF-KURE19 CAR-T Cell Dose
  Participants less than 50 kg:
  * Level -1: 6.5 x 10^6 UF-KURE19 CAR-T Cell Dose
  * Level 1: 11.5 x 10^6 UF-KURE19 CAR-T Cell Dose
  Interventions: Biological: UF-KURE19 CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: UF-KURE19 CAR-T cells — UF-KURE19 cells are initially generated from a starting autologous apheresis sample. T cells are activated and transduced with Kure19 lentiviral vector that consists of a 3rd generation vector with an scFV (FMC63) that targets CD19. The product is harvested at 17-20hr after culture and cryopreserved
Drug: Fludarabine — Fludarabine phosphate is rapidly dephosphorylated to 2-fluoro-ara-A and then phosphorylated intracellularly by deoxycytidine kinase to the active triphosphate, 2-fluoro-ara-ATP. This metabolite appears to act by inhibiting DNA polymerase alpha, ribonucleotide reductase and DNA primase, thus inhibiting DNA synthesis.
  Other Names: Fludara®; Fludarabine Phosphate
Drug: Cyclophosphamide — The mechanism of action is thought to involve cross-linking of tumor cell DNA
  Other Names: Cytoxan ®; Endoxan®; Neosar®; Procytox®; Revimmune®; Cycloblastin®

SUMMARY:
This study seeks to determine the safety and efficacy of the infusion of autologous CD19 CAR-T cells that are manufactured using an ultra-fast process.

DETAILED DESCRIPTION:
This treatment uses T cells already present in the participant's body that have been modified outside of the body by a lentivirus and then returned by an infusion to target the cancer. Lentivirus is a family of viruses that can be used by scientists to alter cells. The specific type of cells that will be used is called UF-KURE19 chimeric antigen receptor T cells (CAR-T cells). The CAR-T cells that will be reinfused into the body are modified using a lentivirus that is no longer active. The investigators are evaluating UF-KURE19 because it uses a process that is shorter than other approved CAR-T cells. While the shorter manufacture time can be an advantage, the safety of this approach has not been demonstrated.

ELIGIBILITY:
Phase 1 Cohort:

Inclusion Criteria:

* Male or female patients aged 18 years or older.
* Participants must have histologically confirmed, CD19 positive (by IHC or flow cytometry) NHL that meets at least one of the following treatment indications.

  * Relapsed after 2 or more lines of chemotherapy, (or)
  * Refractory to chemotherapy, defined as: Progressive disease while receiving last chemotherapy, or Persistent disease after first line chemotherapy treatment with curative intent or stable disease lasting ≤6 months after last chemotherapy, or relapse within 6 months of last chemotherapy, or disease progression or relapse ≤12 months after prior autologous stem cell transplant, (or)
  * Relapsed disease that is ineligible to receive hematopoietic stem cell transplantation due to comorbidities or age or patient preference.
* ECOG Performance status ≤ 2.
* At least one measurable lesion according to Lugano Revised Response Criteria for Malignant Lymphoma.
* Minimum of 2 weeks since prior radiation therapy or systemic therapy to treat malignancy at the time of leukapheresis.
* Total bilirubin ≤ 1.5X institutional upper limit of normal.
* AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal.
* Calculated creatinine clearance ≥ 30mL/min estimated by the Cockcroft - Gault formula.
* Cardiac ejection fraction of ≥45%, and no more than trivial (or trace, minimal or mild) pericardial effusion, as determined by an echocardiogram.
* Adequate pulmonary function, defined as ≤ Grade 1 dyspnea (unless considered secondary to lymphoma) and oxygen saturation (SaO2) ≥ 92% on room air. If pulmonary function tests (PFTs) are performed based on the clinical judgment of the treating physician, patients with forced expiratory volume in 1 second (FEV1)

  ≥ 50% of predicted and diffusing capacity for carbon monoxide (DLCO) (corrected for hemoglobin) of ≥ 40% of predicted will be eligible.
* Participants (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 90 days after the UF-KURE19 CAR-T cell infusion. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.

Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

- For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

* With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the UF-KURE19 CAR-T cell infusion. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the UF-KURE19 CAR-T cell infusion to avoid potential embryonal or fetal exposure.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

* Autologous stem cell transplant within 6 weeks of informed consent.
* History of allogeneic hematopoietic stem cell transplantation.
* Active central nervous system or leptomeningeal involvement by lymphoma. Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal CASE 2422 Page 37 Version 13 02.03.2025 involvement must be in a documented remission by CSF evaluation and contrastenhanced MRI imaging for at least 90 days prior to registration.
* Second active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast).
* Less than 28 days elapsed between prior treatment with investigational agent(s) and leukapheresis.
* New York Heart Association class III-IV congestive heart failure. Cardiovascular disorders including unstable angina pectoris, clinically significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack, or other ischemic event) within 6 months prior to registration.
* Known human immunodeficiency virus infection or acquired immunodeficiency syndrome related illness.
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Evidence of myelodysplastic syndrome or cytogenetic abnormality indicative of myelodysplasia on the most recent bone marrow biopsy prior to initiation of therapy.
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded).
* Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* History of active autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of systemic immunosuppressive medications other than low dose steroids [i.e. maximum of 15mg prednisone equivalent] within the last 6 months.
* Circulating malignant B cells in peripheral blood detected by complete blood count at the time of subject enrollment.

Phase Ib Cohort 1

Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be eligible for enrollment:

* Male or female patients aged 18 years or older.
* Participants must have histologically confirmed, CD19 positive (by IHC or flow cytometry) NHL that meets at least one of the following treatment indications AND there will be a preference for subjects with LBCL including: Diffuse large B-cell lymphoma (DLBCL) not otherwise specified (including DLBCL arising from indolent lymphoma), high-grade B-cell lymphoma, primary mediastinal large B-cell lymphoma, and follicular lymphoma grade 3B.

  * Relapsed after 2 or more lines of chemotherapy, (Or)
  * Refractory to chemotherapy, defined as: Progressive disease while receiving last chemotherapy, or Persistent disease after first line chemotherapy treatment with curative intent or stable disease lasting ≤6 months after last chemotherapy, or relapse within 6 months of last chemotherapy, or disease progression or relapse ≤12 months after prior autologous stem cell transplant, (Or)
  * Relapsed disease that is ineligible to receive hematopoietic stem cell transplantation due to comorbidities or age or patient preference.
* Participants must exhibit both of the following:

  * Nodal lesion: >= 1.5 cm or Non-nodal lesion: >= 1.0 cm
  * FDG avid disease: Deauville Score of 3, 4, or 5 is required. If Deauville Score of 3, Sponsor must confirm eligibility.
* ECOG Performance status ≤ 2 [See Appendix 1].
* Minimum of 2 weeks since prior radiation therapy or systemic therapy to treat malignancy at the time of leukapheresis.
* Total bilirubin ≤ 1.5X institutional upper limit of normal.
* AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal.
* Calculated creatinine clearance ≥ 30mL/min estimated by the Cockcroft - Gault formula. Cardiac ejection fraction of ≥45%, and no more than trivial (or trace, minimal or mild) pericardial effusion, as determined by an echocardiogram.
* Adequate pulmonary function, defined as ≤ Grade 1 dyspnea (unless considered secondary to lymphoma) and oxygen saturation (SaO2) ≥ 92% on room air. If pulmonary function tests (PFTs) are performed based on the clinical judgment of the treating physician, patients with forced expiratory volume in 1 second (FEV1)

  ≥ 50% of predicted and diffusing capacity for carbon monoxide (DLCO) (corrected for hemoglobin) of ≥ 40% of predicted will be eligible.
* Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 90 days after the UF-KURE19 CAR-T cell infusion. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the UF-KURE19 CAR-T cell infusion. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the UF-KURE19 CAR-T cell infusion to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

* Autologous stem cell transplant within 6 weeks of informed consent.
* History of allogeneic hematopoietic stem cell transplantation.
* Active central nervous system or leptomeningeal involvement by lymphoma. Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by CSF evaluation and contrast enhanced MRI imaging for at least 90 days prior to registration.
* Second active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast).
* Less than 28 days elapsed between prior treatment with investigational agent(s) and leukapheresis.
* New York Heart Association class III-IV congestive heart failure.
* Cardiovascular disorders including unstable angina pectoris, clinically significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack, or other ischemic event) within 6 months prior to registration.
* Known human immunodeficiency virus infection or acquired immunodeficiency syndrome related illness. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Evidence of myelodysplastic syndrome or cytogenetic abnormality indicative of myelodysplasia on the most recent bone marrow biopsy prior to initiation of therapy.
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded).
* Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* History of active autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of systemic immunosuppressive medications other than low dose steroids [i.e. maximum of 15mg prednisone equivalent] within the last 6 months.
* Circulating malignant B cells in peripheral blood detected by complete blood count at the time of subject enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Recommended dose(s) of UF-KURE19 CAR-T Cells | Up to 28 days after treatment
  Safety will be assessed by the number of DLT experienced at the target dose which is hypothesized to be less than 33%.
Phase 1: Toxicities associated with the target dose of UF-KURE19 CAR-T Cells | Up to 12 months after treatment
  Toxicities will be reported as specific adverse events as a result of the target dose of UF-KURE19 CAR-T Cells. An adverse event (AE) is any unfavorable or unintended event, physical or psychological, associated with a research study, which causes harm or injury to a research participant as a result of the participant's involvement in a research study.
Phase 1b: Toxicities associated with the target dose of UFKURE19 in patients with Relapsed or Refractory Large B-cell Lymphoma (LBCL). | Up to 12 months after treatment
Phase 1b: Complete response rate (CRR) with UF-KURE19 in patients with Relapsed or Refractory LBCL. | Up to 12 months after treatment
Phase 1b: Objective response rate (ORR, CR + PR) with UF-KURE19 in patients with Relapsed or Refractory LBCL. | Up to 12 months after treatment
Phase 1b: CRR in double/triple hit lymphoma (DHL/THL) patients treated with first-line standard of care chemoimmunotherapy PLUS early intervention of UFKURE19. | Up to 12 months after treatment

SECONDARY OUTCOMES:
Phase 1: Success rate of semi-automated CAR-T manufacturing process | Up to 2 weeks after culture of UF-KURE19 CAR-T cells
  Defined as the percentage of UF-Kure19 CAR-T patient products manufactured that meet the release criteria.
Phase 1: Objective response rates per Lugano Revised Response Criteria for Malignant Lymphoma after treatment with UF-KURE19 in patients with relapsed or refractory non-Hodgkin lymphoma | Up to 12 months after treatment
Phase 1: Complete response rates per Lugano Revised Response Criteria for Malignant Lymphoma after treatment with UF-KURE19 in patients with relapsed or refractory non-Hodgkin lymphoma | Up to 12 months after treatment
Phase 1b cohort of Relapsed or Refractory LBCL: duration of response in patients treated with UF-KURE19 | Up to 12 months after treatment
Phase 1b cohort of Relapsed or Refractory Large B cell Lymphoma(LBCL): Overall survival in patients treated with UF-KURE19 | Up to 12 months after treatment
Phase 1b cohort of Relapsed or Refractory LBCL: Progression-free survival in patients treated with UF-KURE19 | Up to 12 months after treatment
Phase 1b cohort of Relapsed or Refractory LBCL: Manufacturing success rate | Up to 2 weeks after culture of UF-KURE19 CAR-T cells
Phase 1b cohort of DHL/THL: PFS in DHL/THL patients treated with first-line standard of care chemoimmunotherapy PLUS early intervention of UF-KURE19. | Up to 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Changchun Deng, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No